CLINICAL TRIAL: NCT03452319
Title: Effekt av ökad Fysisk träning i Samband Med Thorakoabdominell Esofaguskirurgi
Brief Title: Effects of Increased Physical Activity Before Thoracoabdominal Esophageal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FoU VGR: 238651
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Oesophageal Cancer
Keywords: Thoracoabdominal surgery; Physical Therapy; Inspiratory Muscle Training; Physical Activity
MeSH Terms: conditions — Esophageal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: A single blind, randomized, controlled, intervention study. Evaluation of the addition of increased physical activity and respiratory muscle training for patients undergoing thoracoabdominal esophagus resection compared to standard care
Who Masked: Investigator
Masking Description: Assessor will not be aware of which group the patients are included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pretraining (Experimental): Increased physical activity daily Daily strength training Daily inspiratory and expiratory muscle training Standard care during hospital stay and continued training after discharge.
  Interventions: Other: Pretraining
- Usual care treatment (Active Comparator): Standard care including preoperative information and postoperative breathing exercises and mobilization during hospital stay.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pretraining — Increased physical activity, and daily strength training and breathing exercises.
  Arms: Pretraining
Other: Usual care — Preoperative information
  Arms: Usual care treatment

SUMMARY:
Thoracoabdominal oesophageal resection for cancer is a procedure with high risks for complications, and patients' preoperative status is a crucial factor for outcome. There are only a few studies that evaluate the effect of preoperative intervention, including physical exercises and breathing exercises, after this type of surgery.

The aim of the study is therefore to evaluate the effect of a training intervention before resection of the oesophagus.

One hundred patients scheduled for oesophagus resection according to Ivor-Lewis from five different hospitals in Sweden will be included. The patients will be randomized to an intervention group or a control group. The training intervention starts directly after preoperative radiotherapy and chemotherapy are given and lasts until three months postoperatively.

Intervention includes increased physical activity, strength training and respiratory muscle training.

At inclusion and three months after discharge, the patients will undergo tests of physical function and lung function. In addition, they will fill in questionnaires concerning level of physical function, level of physical activity and quality of life. These questionnaires will also be answered one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo thoracoabdominal oesophagus resection at one of the five included centra

Exclusion Criteria:

* < two weeks between inclusion and surgery
* benign reason for surgery
* difficulties in speaking and reading Swedish
* other injury or disease limiting the ability to perform the intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | From inclusion to 3 months postoperatively
  Test of physical capacity

OTHER OUTCOMES:
Spirometry | From inclusion to 3 months postoperatively
  Vital capacity
Respiratory muscle strength | From inclusion to 3 months postoperatively
  Maximal Inspiratory Pressure and maximal expiratory pressure
Hand strength | From inclusion to 3 months postoperatively
  Hand strength (Jamar)
Leg strength- calf strength | From inclusion to 3 months postoperatively
  Heel rise test
Leg strength | From inclusion to 3 months postoperatively
  Chair stands test
Rib cage range of motion | From inclusion to 3 months postoperatively
  Chest excursion and Respiratory Movement Measurement Instrument
Level of physical activity | From inclusion to 1 year postoperatively (The whole study period)
  Scale by Grimby and Frändin
Physical function | From inclusion to 1 year postoperatively (The whole study period)
  Disability Rating Index
Postoperative recovery | From surgery to 1 year postoperatively
  The Postoperative Recovery Profile
Pain in the ribcage | From inclusion to 1 year postoperatively (The whole study period)
  Numeric rating scale, Scale from 0-10 where 0 indicates no pain and 10 worst imaginable pain
Generic Quality of life | From inclusion to 1 year postoperatively (The whole study period)
  EORTC 3 modules

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, phD, Principal Investigator — Sahlgrenska Academy at Gothenburg university, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fagevik Olsen M, Lothgren S, Trolle U, Elf E, Toomvali-Petersson S, Hermansson M, Hammerlid E, Smedh U. Positive effects of a perioperative training intervention in Ivor Lewis oesophageal surgery: a randomised, controlled multicentre trial. BMC Surg. 2025 Dec 11;26(1):34. doi: 10.1186/s12893-025-03416-4. PMID 41372748